CLINICAL TRIAL: NCT03415620
Title: The Use of Perioperative Music Listening on Anxiety, Pain, Analgesia Use and Patient Satisfaction in Patients Undergoing Surgery
Brief Title: Perioperative Music Listening on Anxiety, Pain, Analgesia Use and Patient Satisfaction
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: KK Women's and Children's Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MT2017-01
Record Dates: First submitted 2018-01-10; First posted 2018-01-30 (Actual); Last update posted 2024-10-10 (Actual); Status verified 2024-10

CONDITIONS: Music; Pain; Anxiety; Patient Satisfaction; Analgesia
MeSH Terms: conditions — Pain; Anxiety Disorders; Patient Satisfaction; Agnosia

STUDY DESIGN:
Intervention Model Description: The randomized controlled phase will recruit 110 parturients.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Music listening (Experimental): Phase 1: Before and after surgery, 300 patients will be offered an ipod with earphone, in which the ipod is equipped with saved playlist of different music genres to select from pre-determined lists of music of different genres or patient choice. Patient will choose the desired playlist and listen to the music for about 30 minutes. Hospital Anxiety and Depression Scale (HADS) score, pain scores, analgesia usage, patient satisfaction, and quality of life measurement will be collected. Analysis of the type of music, duration of music listening, and the genre chosen will be analysed.
  Phase 2: One hundred and ten women undergoing Caesarean delivery assigned to experimental (music listening) group will listen to the music before, during and after surgery. Pain and psychological assessments and demographic data collection will be conducted before and after surgery.
  Interventions: Procedure: Music listening
- No Music Listening (No Intervention): Phase 2: Patients assigned to this group (n=55) will only have pain, psychological assessments and demographic data collection conducted before and after surgery.

INTERVENTIONS:
Procedure: Music listening — Patient is given an ipod with earphone and with saved playlist of different music genres. Music listening session will be given for 30 minutes before, during and after surgery. Questionnaires will be asked to fill in. All the earphones will be disinfected following the hospital's infection control guideline.
  Arms: Music listening

SUMMARY:
The use of music to relieve pain has been studied in many forms of medicines and has been proven to reduce anxiety, pain and analgesic use in the perioperative setting. However, music listening as an inexpensive and duplicable method has not been investigated and implemented in the local context. The investigators hereby propose a prospective study to recruit patients undergoing surgery to evaluate the effectiveness of music in pain relief and post-operative recovery; as well as the implementation and operational readiness of music listening.

DETAILED DESCRIPTION:
Some tissue injury is often unavoidable during surgery, which leads to unavoidable pain and anxiety during the perioperative and post-operative period. Acute post-operative pain and anxiety have been managed via pharmacological interventions. However, non-pharmacological interventions have also been shown to be safe and cost-effective, improve the overall patient experience, and improve outcomes across a variety of surgical settings.

Music has been shown to decrease perioperative pain and modulate the inflammatory response. Additionally, anxiety scores and pain scores have shown statistically significant reductions in the perioperative period, when music therapy was available. Currently only few studies investigate its effects during perioperative period especially in local setting. Thus, the investigators will investigate the feasibility and practicability of deploying music listening in KKH pain management and further determine the nature of the music (duration, genre) by fitting the local context in order to improve the patient outcome in perioperative settings.

Phase 1: A total of 300 patients will be offered to select from pre-determined lists of music of different genres or patient choice, before and after surgery. Hospital Anxiety and Depression Scale (HADS) score, pain scores, analgesia usage, patient satisfaction, and quality of life measurement will be collected. Analysis of the type of music, duration of music listening, and the genre chosen will be analysed.

Phase 2: A hundred and ten women undergoing Caesarean delivery at KK Women's and Children's Hospital (KKH) in 1:1 allocation ratio of experimental (music listening) and control (no music listening) groups. Pain and psychological assessments and demographic data collection will be conducted before surgery, and those allocated to experimental group will be asked to use music listening before, during and after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Healthy participants who are American Society of Anesthesiologists (ASA) 1 and 2 (with well-controlled medical problems);
* Undergo day surgery, same-day-admission gynecologic surgery or cesarean section;
* No hearing impairment.

Exclusion Criteria:

* Patients with significant respiratory disease and obstructive sleep apnea;
* Patients who are unable to read and understand the hospital anxiety questionnaire.

Ages: 21 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Only females undergoing gynecologic surgery or cesarean section in KKH will be recruited.
Enrollment: 410 (Estimated)
Dates: Start 2018-01-03 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Pain score | Baseline and 1 day
  Difference of Pain score before and after surgery. Pain scores (Numeric Rating Scale 0-10) will be asked, with zero being no pain, and 10 being the worst pain possible.

SECONDARY OUTCOMES:
Change in Analgesia usage | Baseline and 1 day
  Analgesia usage (name and dosage of pain medication) used before and after surgery
Change in Patient's satisfaction with the use of music listening (only music listening group) | Baseline and 1 day
  Patient's satisfaction on music listening before and after surgery. Patient will be asked on their satisfaction level based on ordinal scale (Excellent, Good, Fair, Poor).
Change in Hospital Anxiety and Depression Scale (HADS) score (Phase 1 only) | Baseline and 1 day
  HADS Anxiety and Depression score before and after surgery. HADS is commonly used by doctors to determine the levels of anxiety and depression that a patient is experiencing. Each item on the questionnaire is scored from 0-3 and this means that a person can score between 0 and 21 for either anxiety or depression. The HADS uses a scale and therefore the data returned from the HADS is ordinal. For each subscore (anxiety/depression), 0-7 = Normal; 8-10 = Borderline abnormal (borderline case); and 11-21 = Abnormal (case).
Change in EQ-5D-3L score | Baseline and 1 day
  EQ-5D-3L score before and after surgery. EQ-5D-3L is a standardized instrument for measuring generic health status. It is made up for two components; health state description and evaluation. The health status is measured in terms of five dimensions (5D); mobility, self-care, usual activities, pain/discomfort, and anxiety/depression; each dimension ranging from 1-3. From these five dimensions, EQ-5D index is calculated, having a value between 0-1. The evaluation part involves an analogue scale, asking to mark health status on the day of the interview on a 20 cm vertical scale with end points of 0 and 100. Zero corresponds to " the worst health you can imagine", and hundred corresponds to "the best health you can imagine".
Change in Visual analog scale - anxiety (VAS-A) score | Baseline and 1 day
  VAS-A score before and after surgery. A visual analogue scale depicting anxiety (VAS-A) comprises a 10 cm line will be administered, on which the participant marks her current degree of anxiety with the left end of the line being labelled "no anxiety" and the right end being labelled "maximum anxiety".

CONTACTS AND LOCATIONS:
Overall Officials: Ban Leong Sng, MBBS, MMED, Principal Investigator — KK Women's and Children's Hospital
Locations (1):
- KK Women's and Children's Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kakde A, Lim MJ, Shen H, Tan HS, Tan CW, Sultana R, Sng BL. Effect of music listening on perioperative anxiety, acute pain and pain catastrophizing in women undergoing elective cesarean delivery: a randomized controlled trial. BMC Anesthesiol. 2023 Apr 3;23(1):109. doi: 10.1186/s12871-023-02060-w. PMID 37013499